CLINICAL TRIAL: NCT03521492
Title: The Relationship Between Vitamin D Status and Early Childhood Caries Development: A Case-Control Piolet Study
Brief Title: Vitamin D Status With Early Childhood Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Ghazi S. AlAnazi, Pedodontist, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Serum Vitamin D Level
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Early Childhood Caries, Vitamin D Deficiency
Keywords: Early childhood caries, Vitamin D deficiency, Parathyroid hormone, Calcium
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caries group (Experimental)
  Interventions: Diagnostic Test: serum vitamin D , calcium , parathyroid hormone and albumin level
- free caries group (Experimental)
  Interventions: Diagnostic Test: serum vitamin D , calcium , parathyroid hormone and albumin level

INTERVENTIONS:
Diagnostic Test: serum vitamin D , calcium , parathyroid hormone and albumin level — measuring serum level of Vit. D, PTH, Calcium, and Albumin levels

SUMMARY:
Studies that give people vitamin D supplements to prevent caries have found that vitamin D is effective at preventing the development of caries.

The aim of Study:

To determine if there is a relationship between vitamin D deficiency and the development of Early Childhood Caries (ECC).

DETAILED DESCRIPTION:
Methodology:

This is a case-control pilot study to determine the relationship of vitamin D deficiency to the prevalence and severity of ECC. Patient selection and examination following inclusion and exclusion criteria, an Informed consent form will obtain from the parent or guardian after explaining the study in detail. Patients have a yearly pediatric medicine exam and blood drawn regardless of their participation in the study.

Inclusion Criteria:

* Cases: Patients diagnosed with ECC who are treatment planned to receive full mouth dental rehabilitation under General Anesthesia (GA).
* Age 71 months or younger.
* Patients with an American Society of Anesthesiologists (ASA) Classification of 1 (Healthy person).
* Controls: patients who present with no frank cavitated lesions upon visual and radiographic examination who are:
* Patients of record at SFH for an annual exam with blood work patients will schedule to undergo an otolaryngology procedure under GA.

Exclusion Criteria:

* Patients with significant metabolic disorders and/or complex medical issues.
* Patients with an ASA Classification of 2 or greater.
* Patients received vitamin D supply
* Controls: patients who present with frank cavitated lesions upon visual and radiographic examination.

Blood Samples:

The operating room (OR) staff obtained blood samples while the patient will be under GA prior to the initiation of dental treatment. An intravenous (IV) line will place while the child is in the OR for clinical purposes. No additional needle sticks will incur, as blood will draw from a clinically necessary IV line. The sample will obtain as a maximum fill of a Red topped 4.0 mL BD Vacutainer tube. Patients will assign a Research Medical Record Number in the Center Hospital database so that blood samples are correctly will analyze and tabulate when they will leave the OR. Phlebotomist obtained blood from the caries free controls, a topical anesthetic (EMLA) was applied to the antecubital fossa one hour prior to minimize discomfort from the venipuncture during their annual exams also assigned a research related identification number in the same manner.

Vitamin D Analyses:

All blood samples were analyzed for 25-OH Vitamin D levels, PTH level, Ca level and Albumin in Medical Laboratory. Total 25-OH Vitamin D was calculated as the sum total of 25-OH Vitamin D3 and 25-OH Vitamin D2. Lab results were entered into a database and chart for data analysis. PTH, Albumin and Ca levels were analyzed with the same blood sample in addition to 25(OH) D levels. PTH is a more sensitive surrogate for mild Vitamin D deficiency and is typically was analyzed in conjunction with Vitamin D. Analysis and report data are based on the following values: Deficient (< 35 nmol/L), Adequate (≥ 50 nmol/L), Optimal (≥ 75 nmol/L). Normal reference ranges were adopted for calcium (2.1-2.6 mmol/L), albumin (35-47 g/L for those < 48 months and 33-39 g/L for those ≥ 48 months), and PTH (7-50 ng/L). Blood work drawn was analyzed and any discrepancy in findings, such as vitamin D deficiency, was reported to the patient so that they will referrer for treatment by their pediatrician.

Statistical Analysis:

Analysis included descriptive statistics (frequencies, means ± Standard Deviations (SD)), Chi-square analysis, and t-tests. Unadjusted odds ratios (OR) and 95% confidence intervals (CI) were also calculated. Multiple regression analysis was performed for mean 25(OH)D including independent variables significantly associated with vitamin D levels on bivariate analysis or known to influence vitamin D status. Logistic regression for S-ECC including variables associated at the bivariate level was also performed. In both models, some variables were excluded when there was evidence of multi-colinearity. A p value ≤ 0.05 was significant. All analyses will be done by using SPSS 20 software at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Patients diagnosed with ECC who are treatment planned to receive full mouth dental rehabilitation under General Anesthesia (GA).
* Age 71 months or younger.
* Patients with an American Society of Anesthesiologists (ASA) Classification of 1 (Healthy person).
* Controls: patients who present with no frank cavitated lesions upon visual and radiographic examination who are:
* Patients of record at SFH for an annual exam with blood work patients will schedule to undergo an otolaryngology procedure under GA.

Exclusion Criteria:

Exclusion Criteria:

* Patients with significant metabolic disorders and/or complex medical issues.
* Patients with an ASA Classification of 2 or greater.
* Patients received vitamin D supply
* Controls: patients who present with frank cavitated lesions upon visual and radiographic examination.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
vitamin D level of caries and caries free groups | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Ghazi S. Alenazi, MSC, Principal Investigator — M.O.H.
Locations (1):
- Reem Al-Nathsha, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schroth RJ, Levi JA, Sellers EA, Friel J, Kliewer E, Moffatt ME. Vitamin D status of children with severe early childhood caries: a case-control study. BMC Pediatr. 2013 Oct 25;13:174. doi: 10.1186/1471-2431-13-174. PMID 24160554
- [Result] Schroth RJ, Jeal NS, Kliewer E, Sellers EA. The relationship between vitamin D and severe early childhood caries: a pilot study. Int J Vitam Nutr Res. 2012 Feb;82(1):53-62. doi: 10.1024/0300-9831/a000094. PMID 22811377
- [Result] Schroth RJ, Lavelle C, Tate R, Bruce S, Billings RJ, Moffatt ME. Prenatal vitamin D and dental caries in infants. Pediatrics. 2014 May;133(5):e1277-84. doi: 10.1542/peds.2013-2215. PMID 24753535
- [Result] Schroth RJ, Rabbani R, Loewen G, Moffatt ME. Vitamin D and Dental Caries in Children. J Dent Res. 2016 Feb;95(2):173-9. doi: 10.1177/0022034515616335. Epub 2015 Nov 9. PMID 26553883
- [Result] Wojcik D, Krzewska A, Szalewski L, Pietryka-Michalowska E, Szalewska M, Krzewski S, Pels E, Ben-Skowronek I. Dental caries and vitamin D3 in children with growth hormone deficiency: A STROBE compliant study. Medicine (Baltimore). 2018 Feb;97(8):e9811. doi: 10.1097/MD.0000000000009811. PMID 29465564